CLINICAL TRIAL: NCT01045018
Title: BE Study With Clinical Endpoints Comparing Mesalamine Delayed Release Tablets 400 mg to the Reference Listed Drug ASACOL® Delayed Release Tablets 400 mg in Patients With Mild to Moderately Active Ulcerative Colitis
Brief Title: A BE Study Comparing Mesalamine 400 mg to ASACOL® 400 mg in Patients With Mild To Moderately Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMET Pharmaceuticals, LLC (Industry)
Collaborators: Eagle Pharmaceuticals, Inc. (Industry)
Responsible Party: Steve Roth, Managing Partner, EMET Pharmaceuticals, LLC
Allocation: Randomized | Model: Parallel
Other Study IDs: EMET 001
Record Dates: First submitted 2009-12-17; First posted 2010-01-08 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2009-12

CONDITIONS: Mild to Moderate Ulcerative Colitis
Keywords: colitis; ulcerative; ulcerative colitis
MeSH Terms: conditions — Colitis; Ulcer; Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- mesalamine 400 mg tablet (Active Comparator)
  Interventions: Drug: Mesalamine
- Asacol 400 mg Delayed Release Tablet (Active Comparator)
  Interventions: Drug: Mesalamine
- Placebo delayed release tablet (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — placebo 400 mg
  Arms: Placebo delayed release tablet
Drug: Mesalamine
  Arms: mesalamine 400 mg tablet
Drug: Mesalamine
  Arms: Asacol 400 mg Delayed Release Tablet

SUMMARY:
The objectives of this bioequivalence study in patients with ulcerative colitis (UC) were:

* To establish the therapeutic equivalence of mesalamine delayed release tablet (MDRT) and Asacol Delayed Release Tablets 2.4 g per day (800 mg three times daily) and
* To evaluate the safety of MDRT 2.4 g per day (800 mg three times daily) compared to placebo.

DETAILED DESCRIPTION:
This was a multi-center, randomized, parallel-groups comparison of two mesalamine products for treatment of ulcerative colitis. Patients were randomly assigned in an optimized 2:2:1 ratio to MDRT 2.4 g/day, Asacol 2.4 g/day, or placebo. The study was partially blinded due to the difficulties associated with creating placebo that matched both MDRT and Asacol; the placebo matched the MDRT formulation. Placebo groups served as control in the parallel group comparison between MDRT and Asacol. Patients were treated for 6 weeks after randomization and followed through Day 56, which was considered of sufficient length to accommodate any safety issues and to assess efficacy based upon prior clinical trials of mesalamine in patients with mild to moderate active UC as described in the introduction

ELIGIBILITY:
Inclusion Criteria:

Adults with newly diagnosed ulcerative colitis or with relapse following prior treatment and who met all the following criteria were eligible for participation in the study:

1. IRB approved consent form signed and dated prior to any study-related activities
2. Male or, if female, had undergone sterilization (hysterectomy or bilateral tubal ligation), was post-menopausal (defined as 1 year without menses) or has a negative pregnancy test at screening and, if heterosexually active, had used and agreed to continue to use: double-barrier method of contraception (condom and spermicide), oral or patch contraceptives, intrauterine device, or was in a monogamous relationship with a partner who had undergone a vasectomy.
3. 18 years of age or older
4. Newly diagnosed with ulcerative colitis or relapsed following prior treatment
5. Patient had not taken > 1.6 g/day of mesalamine or equivalent for 14 days prior to randomization
6. Disease extending ≥ 15 cm above the anal verge on screening sigmoidoscopy or colonoscopy with confirming biopsy
7. Mild to moderate ulcerative colitis, defined as a Disease Activity Index (DAI) score between 4 and 9, inclusive, at study entry, and with a PGA of 1 or 2 and mucosal appearance (determined by endoscopy exam) score of 1 or 2 (mild/moderate)
8. Able and willing to have kept a daily diary during the study

Exclusion Criteria:

1. Treatment with topical rectal, oral, or intravenous (IV) corticosteroids within 30 days of screening or immunosuppressives (e.g. azathioprine, 6-mercaptopurine) within the 90 days immediately preceding Screening
2. Use of rectal - administered aminosalicylates within 7 days of randomization
3. Patient had taken greater than 1.6 g/day of mesalamine or equivalent within 14 days of randomization
4. Crohn's disease, ischemic colitis, or disease of bacterial origin
5. Known allergy or hypersensitivity to aspirin or salicylate compounds
6. History of or laboratory results showing significant hepatic or renal disease or other significant medical condition which in the opinion of the investigator precluded participation in the study based on efficacy/safety assessments
7. History of cancer other than basal cell carcinoma within the five years immediately preceding study entry
8. In relapse for > 3 weeks prior to the screening visit
9. Proctitis below 15 cm from the anal verge
10. History of or current gastrointestinal bleeding other than bloody stools associated with ulcerative colitis
11. History of bleeding disorder
12. Active peptic ulcer disease, history of gastrointestinal obstruction including severe constipation, or anatomic abnormality of the GI tract
13. Previous colonic surgery
14. History of alcohol or other substance abuse within the year immediately preceding anticipated study entry
15. HIV positive
16. > 6 bloody stools per day
17. Positive stool culture for ova and/or parasites, enteric pathogens including Salmonella, Shigella, Yersinia, and Campylobacter, or positive stool assay for C. difficile toxin
18. Pregnant or breast feeding
19. Used an investigational drug in the 30 days prior to randomization
20. BUN or serum creatinine levels of 1.5 times the upper limit of normal (ULN) or liver enzyme levels > 2 times the ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Treatment Success: Responders are patients in remission or who do not require use of rescue medication for symptomatic relief of UC at week 6 Treatment benefit: Improvement at endpoint compared to baseline Treatment Failure: Increase or no improvement | 4 months

SECONDARY OUTCOMES:
Tolerability and safety will be determined by evaluation of AEs, SAEs, hematology, serum chemistry and urinalysis | 4 months